CLINICAL TRIAL: NCT01526382
Title: Use of PiCCO System in Critically Ill Patients With Septic Shock and Acute Respiratory
Brief Title: Use of PiCCO System in Critically Ill Patients With Septic Shock and Acute Respiratory Distress Syndrome
Acronym: PiCCO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongheng Zhang, principal investigator, Jinhua Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZZH-01
Record Dates: First submitted 2012-01-27; First posted 2012-02-03 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2012-09

CONDITIONS: Septic Shock; Acute Respiratory Distress Syndrome
Keywords: septic shock; acute respiratory distress syndrome; transpulmonary thermodilution technique; mortality
MeSH Terms: conditions — Shock, Septic; Respiratory Distress Syndrome | interventions — Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- intervention arm (Active Comparator): patients allocated to intervention arm receive PiCCO monitoring for hemodynamics and pulmonary conditions
  Interventions: Device: PiCCO monitoring (PULSION)
- control arm (Placebo Comparator): Patients in this arm do not receive PiCCO monitoring device to guide fluid management, but central venous catheter can be inserted at the discretion of treating physician.
  Interventions: Procedure: central venous catheter

INTERVENTIONS:
Device: PiCCO monitoring (PULSION) — Patients are monitored with PiCCO system.
  Other Names: PiCCO (pulsion medical system, PULSION PiCCO plus)
  Arms: intervention arm
Procedure: central venous catheter — patients in this arm can receive central venous catheter
  Arms: control arm

SUMMARY:
PiCCO has been widely used in critical care settings for several decades. Together with pulmonary artery catheter, it is regarded as the important tool for guiding fluid management in patients with shock or acute respiratory distress syndrome. However, its effects on patients' outcome remain untested. The investigators study is a pilot study that is designed to test whether the use of PiCCO will improve patients' outcome, as compared to those without PiCCO monitoring.

DETAILED DESCRIPTION:
PiCCO comprises techniques of pulse contour analysis and transpulmonary thermodilution, and can provide important information on hemodynamics and pulmonary functions. It has been widely used in critical care settings for several decades. Together with pulmonary artery catheter (PAC), it is regarded as the important tool for guiding fluid management in patients with shock or acute respiratory distress syndrome. During last two decades, many well designed clinical trials have been conducted to see whether the use of PAC would benefit patient outcome. The result consistently showed that PAC added no benefit in terms of mortality, ICU length of stay, organ failure free survival days, and the length of mechanical ventilation. Since PiCCO is relatively new to PAC, and its effects on patients' outcome remain untested. The investigators study is a pilot study that is designed to test whether the use of PiCCO will improve patients' outcome, as compared to those without PiCCO monitoring.

ELIGIBILITY:
Inclusion Criteria:

Patients were included if they were diagnosed with Shock, Acute respiratory distress syndrome (ARDS), or both.

Shock was defined by the presence 4 criteria:

* Heart rate of at least 90/min;
* A respiratory rate of at least 20/min or a PaCO2 of 32mmHg or lower or the use of mechanical ventilation;
* The use of vasopressors to maintain a systolic blood pressure of at least 90mmHg despite fluid resuscitation, low dose of dopamine (≤ 5 μg/kg per minute), or dobutamine;
* at least 1 of 3 signs of hypoperfusion (urine output < 0.5mL/kg of body weight per hour for 1 hour or more; neurologic dysfunction defined by confusion, psychosis, or a Glasgow coma scale score of ≤ 6; plasma lactate higher than the upper limit of the normal value).

Acute respiratory distress syndrome：

* the presence of acute decrease in PaO2/FIO2 to 200mmHg or lower,
* bilateral pulmonary infiltrates or a chest radiograph consistent with edema;
* no clinical evidence of left atrial hypertension; and requirement for positive pressure ventilation.

Exclusion Criteria:

* Patients were moribund.
* signed do-not-resuscitation odor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days
  death from any cause before day 30

SECONDARY OUTCOMES:
14 day mortality | 14 days
  patients were followed up for 14 days
ICU length of stay | up to 30 days
  the time from ICU admission to ICU discharge or death
days on mechanical ventilation | up to 30 days
  days during which the patients are on mechnical ventilation: The criteria for termination of mechanical ventilation: a cooperative patient, recovery from primary disease, hemodynamically stable, adequate and strong cough reflex, positive end-expiratory pressure <5 cmH2O, pressure support <10 cmH2O and the spontaneous breathing trial is successfully passed.
days of vasoactive agents support | up to 30 days
  days during which vasoactive agents are used: The sum of the number of days with one or more vasoactive agents to maintain a mean arterial pressure >60 mmHg
ICU free survival days during 30-day period | 30 days
  ICU free survival days during 30-day period
mechanical ventilation free survival days during 30-day period | 28 days
  mechanical ventilation free survival days during 30-day period

CONTACTS AND LOCATIONS:
Overall Officials: Zhongheng Zhang, MD, Study Chair — Jinhua Municipal Central Hospital
Locations (2):
- China (2):
  - department of critical care medicine, Jinhua central hospital, Jinhua, Zhejiang
  - Traditional Chinese Medical hospital of Jinhua City, Jinhua, Zhejiang

REFERENCES:
- [Background] Richard C, Warszawski J, Anguel N, Deye N, Combes A, Barnoud D, Boulain T, Lefort Y, Fartoukh M, Baud F, Boyer A, Brochard L, Teboul JL; French Pulmonary Artery Catheter Study Group. Early use of the pulmonary artery catheter and outcomes in patients with shock and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2003 Nov 26;290(20):2713-20. doi: 10.1001/jama.290.20.2713. PMID 14645314
- [Derived] Zhang Z, Xu X, Yao M, Chen H, Ni H, Fan H. Use of the PiCCO system in critically ill patients with septic shock and acute respiratory distress syndrome: a study protocol for a randomized controlled trial. Trials. 2013 Feb 1;14:32. doi: 10.1186/1745-6215-14-32. PMID 23374652